CLINICAL TRIAL: NCT02094339
Title: Comparison of Three Kinds of Postoperative Analgesia After Total Knee Arthroplasty :a Randomized Clinical Trial
Brief Title: Comparison of Three Kinds of Postoperative Analgesia After Total Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, bo xu, associate chief physician, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Unilateral Knee Replacement
Record Dates: First submitted 2014-03-19; First posted 2014-03-21 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Pain; Complications
Keywords: Local analgesia system; Ropivacaine; Analgesic efficacy after operation; Postoperative
MeSH Terms: conditions — Pain | interventions — Nerve Block; Ropivacaine; Analgesics, Opioid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Local analgesic (Experimental): This group uses local analgesia infusion pump of 0.2% ropivacaine 360ml through periarticular infiltration for postoperative analgesia.
  Interventions: Procedure: Local analgesic; Drug: ropivacaine
- Nerve Block (Active Comparator): People in this group will receive a postoperative pain management by continuous lumbar plexus block with 0.2% ropivacaine.
  Interventions: Procedure: Nerve Block; Drug: ropivacaine
- Intravenous analgesic (Active Comparator): This group is treated with intravenous electronic analgesia pump infusion of flurbiprofen axetil 250mg,palonosetron 0.5mg,pentazocine 240mg.dezocine 30mg.
  Interventions: Procedure: Intravenous analgesic; Drug: opioid

INTERVENTIONS:
Procedure: Local analgesic — Patient will be performed under combined lumbar plexus and sciatic nerve block with 0.33% ropivacaine.At the end of surgery,two catheters are left in the wound.One is intraarticular and the other is on the surface of articular cavity.And then a pump elastomeric infusion pump will be connected with the catheters, which runs 5mL every hours.
  Arms: Local analgesic
Procedure: Nerve Block — Combined lumbar plexus and sciatic nerve block with 0.33% ropivacaine will be performed before the surgery.After the a bolus of 30mL ropivacaine around lumbar plexus,a catheter will be left in Psoas gap with 6cm.A pump elastomeric infusion pump running 5mL every hours will also be connected with the catheters at the end of the operation.
  Arms: Nerve Block
Procedure: Intravenous analgesic — People in this group will also receive an anesthesia of combined lumbar plexus and sciatic nerve block with 0.33% ropivacaine.An intravenous electronic analgesia pump infusion of flurbiprofen axetil 250mg,palonosetron 0.5mg,pentazocine 240mg.dezocine 30mg will will provide postoperative pain management.The patients will received a 2 mL/h continuous basal infusion and 1 mL boluses with a lockout time of 30 min after a 5 mL Loading dose at the end of the surgery.
  Arms: Intravenous analgesic
Drug: ropivacaine — 0.2% ropivacaine
  Arms: Local analgesic
Drug: ropivacaine — 0.2% ropivacaine
  Arms: Nerve Block
Drug: opioid — flurbiprofen axetil 250mg,palonosetron 0.5mg,pentazocine 240mg.dezocine 30mg
  Arms: Intravenous analgesic

SUMMARY:
Postoperative pain after total knee arthroplasty (TKA) can be difficult to manage and may delay recovery. There are multimodal postoperative pain management after TKA, including intravenous opioids, epidural analgesia, peripheral nerve blocks or periarticular infiltration with local anesthetics. All of these treatments may lead to side effects such as nausea, headache, hypotension, urinary retention, partial motor block and infection of the knee. Therefore the investigators will compare three methods of postoperative analgesic after TKA by their efficiency and complication.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of American Association of anesthetists（ASA）Grade 1、2 or 3
2. Aged between 18 and 85 years
3. Undergoing elective total knee replacement

Exclusion Criteria:

1. Mental illness can not match
2. Nerve block, epidural anesthesia contraindicated
3. People who have Slow-type arrhythmias
4. History of chronic headaches and long-term use of analgesic drugs
5. People who were postoperative consciousness, language or hearing impaired

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
pain | 72 hours postoperation
  Up to 72 hours after operation,postoperative pain visual analogue scale(VAS) scores are used to evaluate the level of pain.

SECONDARY OUTCOMES:
sedation | 72 hours postoperation
  At 2, 4, 6, 12, 24, 36, 48,72 hours after operation,sedation OAA/S scores are used to evaluate the level of sedation.
complication | 72 hours postoperation
  Investigators document the incidence of nausea,vomiting,headache,urinary retention and et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Military Region General Hospital, Department of Anesthesiology, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Toftdahl K, Nikolajsen L, Haraldsted V, Madsen F, Tonnesen EK, Soballe K. Comparison of peri- and intraarticular analgesia with femoral nerve block after total knee arthroplasty: a randomized clinical trial. Acta Orthop. 2007 Apr;78(2):172-9. doi: 10.1080/17453670710013645. PMID 17464603
- [Result] Serpell MG, Millar FA, Thomson MF. Comparison of lumbar plexus block versus conventional opioid analgesia after total knee replacement. Anaesthesia. 1991 Apr;46(4):275-7. doi: 10.1111/j.1365-2044.1991.tb11495.x. PMID 2024744